CLINICAL TRIAL: NCT06278636
Title: Laparoscopic Ultrasound Examination: Analysis of Feasibility and fEllows Surgeons' LEarning Curve in Minimally Invasive Gynecological Procedures
Brief Title: Laparoscopic Ultrasound Examination: Analysis of Feasibility
Acronym: LUXA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mascilini Floriana, Ph.D, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5745
Record Dates: First submitted 2023-06-23; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-06

CONDITIONS: Gynecologic Cancer; Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laparoscopi ultrasound examination — Analysis of feasibility and fellow surgeons learning curve in minimally invasive gynecological procedures

SUMMARY:
This is a prospective cohort study to assess the feasibility of the laparoscopic ultrasound examination, directly by surgeons, during minimally invasive gynaecological surgery.

The secondary aims are to examine the learning curve for laparoscopic ultrasound examination and the performance score in obtaining high quality ultrasound images of anatomical parameters by a team of 5 gynecological laparoscopic fellows. The patients' medical history and symptoms will also be recorded to define whether these clinical data can influence the failure rate. With advanced technology, the conventional workflow can be simplified by using laparoscopic ultrasound probes directly by surgeons, to utilize the hospital resources efficiently and to reduce operating times. In this regard, we would like to demonstrate that the application of laparoscopic examination is feasible and easy to learn by surgeons. This innovative technique could open up multiple diagnostic and therapeutic opportunities for the patient, providing potential clinical information useful to the surgeon.

DETAILED DESCRIPTION:
The use of laparoscopic ultrasound is an evolving field with a potentially wide range of advantages that could facilitate complex gynecologic surgical procedures; increasing surgical safety by allowing the surgeon to see beyond the surface of the organ, visualizing anatomical structures and identifying, for example, retroperitoneal recurrences and benign or malignant pelvic lesions, even small and not visible laparoscopically, and consequently improving the surgical accuracy of tumor resection. (10) Gynecologists who are familiar with gynecological transvaginal ultrasound should be able to become proficient in identifying pelvic organs during surgical procedures in order to improve surgical accuracy, reduce complications, and ultimately improve patient care.

Nevertheless, this technique has been slow to be implemented in the clinical setting, perhaps due to the lack of a learning curve. Therefore, training gynecological surgical fellows in recognizing pelvic structures using laparoscopic probes is critical for allows them to use this tool in different application fields, providing them with an important advantage. The training of gynecological surgeons in the use of laparoscopic probes would provide an advantage in terms of surgical time, speeding up the procedures of recognition and removal of target lesions. In addition, by making surgeons autonomous in the operating theatre, the need for an additional ultrasound operator during surgery would be eliminated. These benefits would translate into a potential reduction in cost as well

ELIGIBILITY:
Inclusion Criteria:

* Fellow surgeons with EFSUMB level 1 experience of ultrasound in gynecology.
* Women affected by gynecological pathologies undergoing elective laparoscopic surgery such as endometrial cancer, cervical cancer at early stage, or benign pathologies.
* All women will be required to sign written informed consent to enter the study.

Exclusion Criteria:

* Patients affected by gynaecological pathologies undergoing emergency surgeries.
* Refusal to sign written informed consent.
* Patients with previous hysterectomy or salpingo-oophorectomy.
* Uterus and adnexa not visualised at LPS examination.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible population includes 5 fellow surgeons with EFSUMB level 1 experience of ultrasound in gynecology (11) and 150 women satisfying inclusion criteria
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
feasibility of the laparoscopic | 2 minutes
  for to assess the feasibility of the laparoscopic ultrasound examination during minimally invasive gynaecological surgery, achievement of one ultrasound picture in maximum 120 seconds examination during minimally invasive gynaecological surgery, in terms of achievement of one ultrasound picture in maximum 120 seconds

SECONDARY OUTCOMES:
the learning curve of fellow surgeons | 5 minutes
  To investigate the learning curve of fellow surgeons in obtaining skill competency by using laparoscopic probe
the performance of fellow surgeons | 30 minutes
  To evaluate the performance of fellow surgeons in obtaining high-quality US images of anatomical parameters using expert assessment as the gold standard and in achieving a reduction in the operative time of laparoscopic probe use.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Laparoscopic Ultrasound examination: analysis of Feasibility and fEllows Surgeons' LEarning Curve in minimally invasive gynecological procedures